CLINICAL TRIAL: NCT02945813
Title: SAKK 08/15 - PROMET - Multicenter, Randomized Phase II Trial of Salvage Radiotherapy +/- Metformin for Patients With Prostate Cancer After Prostatectomy
Brief Title: SAKK 08/15 - PROMET - Salvage Radiotherapy +/- Metformin for Patients With Prostate Cancer After Prostatectomy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial was prematurely closed for accrual by the SAKK Board and the follow-up period shortened to one year after last RT fraction of the last patient
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAKK 08/15 - PROMET; 2016-003599-39 (EudraCT Number)
Record Dates: First submitted 2016-10-25; First posted 2016-10-26 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Prostate Cancer after Prostatectomy; Phase II Trial; Salvage Radiotherapy; Metformin
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Metformin (Experimental): * Metformin - 850mg PO BID; 48 weeks
  * Salvage radiotherapy SRT - 35 x 2Gy; 7 weeks
  Interventions: Drug: Metformin; Radiation: Salvage Radiotherapy SRT
- Arm B: Salvage Radiotherapy (Active Comparator): - Salvage radiotherapy SRT - 35 x 2Gy; 7 weeks
  Interventions: Radiation: Salvage Radiotherapy SRT

INTERVENTIONS:
Drug: Metformin — 850mg PO BID; 48 weeks
  Arms: Arm A: Metformin
Radiation: Salvage Radiotherapy SRT — SRT 35 x 2Gy; 7 weeks

SUMMARY:
The main objective of the trial is to explore the efficacy of salvage radiotherapy (SRT) plus metformin compared to SRT in the endpoint of time to progression after prostatectomy failure.

DETAILED DESCRIPTION:
Although the use of salvage radiotherapy (SRT) is the only potentially curative treatment after prostatectomy failure, it has provided suboptimal results over the years. Metformin may represent an effective and inexpensive means to improve SRT outcomes with a favorable therapeutic ratio. Taken pre-clinical and retrospective clinical data together, there is a compelling rationale for conducting a RCT with SRT and metformin. Herein we propose a multicenter, randomized, open-label, proof-of-concept phase II trial with the hypothesis that the addition of metformin to SRT can delay time to progression compared to the standard-of-care SRT. The study has 1:1 randomization and stratification variables include Gleason score, PSA at SRT, surgical margin status and ADT use.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to ICH/GCP regulations before registration and prior to any trial specific procedures
* Histologically confirmed adenocarcinoma of the prostate without small cell features
* Tumor stage pT2a-3b, pN0 or cN0, M0, R0-1 resection margins, according to UICC TNM 2009, Gleason score available
* Radical prostatectomy (RP) at least 12 weeks before registration
* PSA progression after RP defined as two consecutive rises with the final PSA > 0.1 ng/mL or three consecutive rises. The first value must be measured earliest 4 weeks after RP
* PSA ≤ 2 ng/mL within 14 days prior to registration
* Age ≥ 18 years at time of registration
* WHO performance status 0-1
* Adequate hepatic function within 14 days prior to registration: bilirubin ≤ 1.5 x ULN (exception if Gilbert's syndrome ≤ 3 x ULN), AST and ALT ≤ 2.5 x ULN
* Adequate renal function within 14 days prior to registration: calculated corrected creatinine clearance ≥ 60 mL/min, according to the formula of corrected Cockcroft-Gault Patient agrees not to father a child and to use effective contraceptive methods during salvage radiotherapy and until 6 months after the last fraction of radiotherapy

Exclusion Criteria:

* Persistent PSA (> 0.4 ng/mL) 4 to 20 weeks after RP
* Pelvic lymph node enlargement > 0.8 cm in short axis diameter (cN positive) assessed by mpMRI within 12 weeks prior to registration, unless the enlarged lymph node is sampled and negative
* Evidence of macroscopic local recurrence assessed by mpMRI within 12 weeks prior to registration
* Palpable prostatic fossa mass suggestive of recurrence, unless an ultrasound guided biopsy is negative for malignancy
* Presence or history of prostate cancer metastases. In case of clinical suspicion (e.g. bone pain), imaging (e.g. bone scan, Choline-PET, PSMA-PET, whole body MRI) must be performed. The imaging method is at the discretion of the investigator.
* If PET/CT scan was performed, any metabolic uptake considered clinically suspicious for malignancy, unless biopsy proves to be negative.
* History of hematologic or primary solid tumor malignancy, unless in remission for at least 3 years from registration with the exception of curatively treated localized non-melanoma skin cancer
* Patients diagnosed with diabetes mellitus
* Treatment with metformin within the last 3 months prior to registration
* Prior pelvic radiotherapy
* Hormonal treatment as bilateral orchiectomy prior or following RP
* Usage of products known to affect PSA levels within 4 weeks prior to start of trial treatment
* Bilateral hip prosthesis
* Severe or active co-morbidity likely to impact on the advisability of salvage RT, e.g.:

  * History of inflammatory bowel disease or any malabsorption syndrome or conditions that would interfere with enteral absorption
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Chronic Obstructive Pulmonary Disease (COPD) exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
* Any condition associated with increased risk of lactic acidosis (e.g. alcohol abuse, congestive heart failure NYHA III or IV
* Clinically significant history of liver disease consistent with Child-Pugh Class B or C, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Severe or uncontrolled kidney disease resulted in impaired kidney function (GFR <60ml/min)
* Any acute or chronic condition that could cause tissue hypoxia (e.g. cardiac or respiratory insufficiency, recent myocardial infarction, shock)
* Treatment with any experimental drug or participation within a clinical trial within 30 days prior to registration (exception: concurrent participation in the biobank project SAKK 63/12 is allowed)
* Any concomitant drug contraindicated for use with metformin according to the approved product information
* Known hypersensitivity to metformin/placebo or to any of its components
* Hereditary intolerance to fructose; known galactose-1-phosphate uridyl transferase deficiency, UDP galactose 4 epimerase deficiency, galactokinase deficiency, Fanconi-Bickel syndrome, congenital lactase deficiency, or glucose-galactose malabsorption (due to the lactose-containing placebo)
* Inability or unwillingness to swallow oral medication
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Time to progression (TTP) | within 18 months after randomization
  The primary endpoint of the trial is time to progression (TTP), defined as time from randomization until one of the following events, whichever comes first:
  * Biochemical progression
  * Clinical progression
  * Death due to clinical progression

SECONDARY OUTCOMES:
Progression free survival (PFS) | within 18 months after randomization
  PFS is defined as time from randomization until one of the following events, whichever comes first:
  * Biochemical progression
  * Clinical progression
  * Death from any cause
Undetectable Prostate Specific Antigen (PSA) under normal testosterone levels | up to 18 months after last radiotherapy fraction
  Undetectable PSA is defined as a serum PSA value of ≤0.05 ng/mL for at least two consecutive measurements after the last radiotherapy fraction and up to 18 months thereafter. To count as undetectable PSA under normal testosterone levels, the testosterone level has to be ≥50 ng/dL (i.e. a non-castrate testosterone level).
50% PSA response | at randomization up to 18 months after last radiotherapy fraction.
  50% PSA response is defined as a ≥50% PSA decline after radiotherapy compared to the serum PSA level at randomization up to 18 months after last radiotherapy fraction.
Clinical progression-free survival | week 64 then every 6 months for the first year and every 12 months thereafter up to 10 years from last RT fraction.
  Clinical progression-free survival will be calculated as the time from randomization until clinical progression or death due to any cause.
Time to further anti-cancer systemic therapy | week 64 then every 6 months for the first year and every 12 months thereafter up to 10 years from last RT fraction.
  Time to further anti-cancer systemic therapy (e.g. hormonal treatment) is defined as the time from randomization to the start of any type of salvage systemic treatment.
Prostate cancer-specific survival (PCSS) | at week 64 then every 6 months for the first year and every 12 months thereafter up to 10 years from last RT fraction.
  Prostate cancer-specific survival will be calculated as the time from randomization to the date of death due to prostate cancer.
Overall survival (OS) | at week 64 then every 6 months for the first year and every 12 months thereafter up to 10 years from last RT fraction.
  Overall survival will be calculated as the time from randomization to the date of death from any cause.
Adverse Events (AE) | until 56 weeks (specific RT-related AEs : until 10 years)
  AEs will be assessed according to NCI CTCAE v4.03.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M. Aebersold, Prof, Study Chair — Bern University Hospital - Radiation Oncology; Alan Dal Pra, MD, Study Chair — Miller School of Medicine, University of Miami
Locations (27):
- France (8):
  - Centre Hospitalier Régional Universitaire (CHRU) Jean Minjoz, Besançon
  - Clinique Pasteur - Centre finistérien de radiothérapie et d'oncologie, Brest
  - Centre de lutte contre le cancer Léon Bérard, Lyon
  - Hôpital Saint-Louis, Paris
  - CHU de Poitiers - La Miletrie, Poitiers
  - Institut de Cancérologie de L'Ouest René Gauducheau, Saint-Herblain
  - Institut de Cancérologie de la Loire Lucien Neuwirth, Saint-Priest-en-Jarez
  - Clinique Pasteur - Oncorad, Toulouse
- Germany (5):
  - Universitätsmedizin Berlin, Berlin
  - Klinikum der Universität München, München
  - Universitätsklinikum Rostock, Rostock
  - Universitätsklinik Tübingen, Tübingen
  - Universitätsklinikum Würzburg, Würzburg
- Switzerland (14):
  - Universitätsspital Basel, Basel
  - EOC-Istituto Oncologico della Svizzera Italiana, Bellinzona
  - Inselspital Bern, Bern
  - Kantonsspital Graubuenden, Chur
  - HFR - Hôpital cantonal, Fribourg
  - Hôpitaux Universitaires Genève HUG, Geneva
  - Clinique de Genolier, Genolier
  - Spital Thurgau, Münsterlingen
  - Kantonsspital St. Gallen, Sankt Gallen
  - Hopital de Sion, Sion
  - Kantonsspital Winterthur, Winterthur
  - Klinik Hirslanden, Zurich
  - Stadtspital Triemli, Zurich
  - UniversitätsSpital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No